CLINICAL TRIAL: NCT02892799
Title: Non-invasive Fluid Management in Critically Ill Patients With ARDS
Brief Title: Non-invasive Fluid Management
Acronym: DECAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Michael Lanspa, Adjunct Assistant Professor, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1050087
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: NICOM device
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care (Active Comparator): Patients randomized to the usual care arm will be treated almost the same as if they do not enroll in the study. They will be managed in accordance with best ICU (intensive care unit) practices, with treatment decisions made by the treating team. Often this will include blood draws (often 2 teaspoons once or twice per day, but sometimes exceeding this), assessments of cardiac function, assessments of fluid status, and other measures as dictated by the presenting illness (this is broad and will include antibiotics, diuretics, cardiac medications, ventilator and oxygen management, etc.). Patients in the usual care arm will not have diuresis managed by NICOM.
  Interventions: Other: Standard of Care
- NICOM-Guided Diuresis (Experimental): Within 4 hours, patients will have their blood pressure obtained, a NICOM-based assessment of PLR (passive leg raise)-induced change in cardiac index, hourly urinary output, and quantization of the total input and output from the beginning of the morning shift (7 am). This will allow determination of the fluid goal over the next 4 hours. Patients will receive furosemide to achieve the goal fluid balance, if needed as described in the accompanying protocol. Monitoring of electrolytes and renal function will be at the discretion of the treating physician.
  Following the initial evaluation, at set times spaced every 4 hours apart, patients will have an ongoing evaluation of the day's fluid balance, hourly urinary output, and PLR/NICOM values. This diuresis protocol will continue for a total of seven 24-hour periods or until the primary means of oxygenation/ventilation has been withdrawn, whichever occurs first. Patients will be followed for a total of 60 days to evaluate outcome data.
  Interventions: Other: NICOM-Guided Diuresis

INTERVENTIONS:
Other: NICOM-Guided Diuresis — NICOM-based assessment of PLR-induced change in cardiac index
  Arms: NICOM-Guided Diuresis
Other: Standard of Care
  Arms: Standard of Care

SUMMARY:
For patients with a condition called acute respiratory distress syndrome (ARDS), managing their fluid levels to achieve a negative balance helps to improve their outcomes. In the past, patients' fluid levels were monitored with central lines placed into the bloodstream. However, most patients are now managed without central lines. A device called a NICOM (noninvasive cardiac output monitor) which monitors patients' heart function, using a few patches which are attached to their chest, may be useful in managing fluid levels without central lines. This study will compare the fluid balance in patients who are managed with typical care to the fluid balance in patients who are managed with the NICOM device.

DETAILED DESCRIPTION:
BACKGROUND:

Negative fluid balance in acute respiratory distress syndrome (ARDS) has been shown to improve intensive care unit (ICU) length of stay and ventilator-free days. Although protocols exist for fluid management, all require invasive hemodynamic monitoring. Despite the large evidence base supporting the use of invasive monitoring, the majority of ARDS patients are now managed without invasive central lines. A non-invasive protocol for managing fluid status in patients with ARDS has not been rigorously implemented nor studied within a randomized controlled trial.

OBJECTIVE:

The study objective is to compare a novel non-invasive parameter-guided protocol for fluid management to usual care. The specific aims are: 1) to compare the incidence of new or worsening renal failure, the incidence of new or worsening shock, and the incidence of new or worsening non-shock hypotension; 2) to compare the relative effectiveness of the 2 treatment groups as assessed by cumulative fluid balance over 7 days; 3) to determine if the non-invasive protocol increases the number of ventilator-free days and ICU-free days; and further, to evaluate if it decreases 60-day mortality; and 4) to document the clinical instances where treatment digression between the 2 groups occurs.

STUDY DESIGN:

This study is a single-blinded, randomized control trial, comparing 1 treatment arm to usual care. We will treat patients with severe hypoxemic respiratory failure (including ARDS) for 7 consecutive days. Their post-study course will be monitored for a period of 60 days or until death. Patients who are randomized to the intervention group will receive fluid management strategies that are dictated by non-invasively derived (via the "NICOM" device) surrogates of cardiac preload and output. Patients who are randomized to the control group will receive standard-of-care "best practice" fluid management, as dictated by the treating physician.

ELIGIBILITY:
Inclusion Criteria

* ≥18 years of age
* Acute respiratory failure (must meet ONE of the following)

  * Receipt of mechanical ventilation
  * Receipt of non-invasive ventilation via BIPAP or CPAP, used for an indication other than sleep apnea
  * Receipt of high flow nasal cannula oxygenation with FiO2 > .4 and a flow rate > 30 LPM
* Increased total body fluid volume (any of the following)

  * > 1 kg increased weight gain (compared to admission)
  * > 1 L positive fluid balance (compared to admission)
  * Bedside clinician determination

Exclusion Criteria

* Known pregnancy (a negative pregnancy test is required for women of child-bearing potential)
* Dialysis dependence, at the time of enrollment
* Chronic ventilator dependence, prior to admission
* Intubation for airway protection (solely for a surgical procedure) or upper airway obstruction
* Neuromuscular disease that impairs the ability to ventilate spontaneously, such as C5 or higher spinal cord injury, amyotrophic lateral sclerosis, Guillain-Barré Syndrome, and myasthenia gravis
* Solid organ transplantation or bone marrow transplantation
* Vasculitis with diffuse alveolar hemorrhage
* Severe chronic liver disease (Child-Pugh Score 10-15)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Composite incidence of new acute kidney injury (AKI), new hypotension (mean arterial blood pressure < 60 following diuresis), and new shock (SOFA (Sequential Organ Failure Assessment) score) | Admission to ICU through discharge from ICU
  Primary predictor is diuresis treatment protocol arm
7-day cumulative fluid balance | Days 1 to 7
  Primary predictor is diuresis treatment protocol arm
Correlation of non-invasive NICOM derived cardiac parameters with incidence of new acute kidney injury (AKI), new hypotension, and new shock | Admission to ICU through discharge from ICU
  Primary predictor is NICOM-derived percent (%) change in stroke volume index

SECONDARY OUTCOMES:
Incidence of new kidney injury | Days 1-7
  New kidney injury is defined by an increase in serum creatinine, adjusted for a fluid balance of 50%, or an absolute increase in serum creatinine of more than 0.3-mg/dL over a 48-hour window during study days 1-7
Ventilator-free days to day 28 (days alive and free from mechanical ventilation) | Admission to ICU to day 28 after admission to ICU
ICU-free days to day 28 (days alive and out of the ICU) | Admission to ICU to day 28 after admission to ICU
60-day mortality | Admission to ICU to 60 days after admission to ICU
Incidence of new shock between the treatment arms (NICOM-guided diuresis, usual care) | Admission to ICU through discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lanspa, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No